CLINICAL TRIAL: NCT01492309
Title: Transcranial Magnetic Stimulation (TMS) in Pregnant Women With Depressive Disorder
Brief Title: Beat the Blues in Pregnancy Study - Transcranial Magnetic Stimulation
Acronym: TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 812494; K23MH092399 (NIH)
Record Dates: First submitted 2011-12-03; First posted 2011-12-14 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Pregnancy; Brain Derived Neurotrophic Factor; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- Active Transcranial Magnetic Stimulation (Active Comparator): 38 pregnant women with MDD will be randomized to receive active 1 Hz right-sided dorsolateral prefrontal cortex (DLPFC) TMS.
  Interventions: Device: Active Transcranial Magnetic Simulation
- Sham Transcranial Magnetic Stimulation (Sham Comparator): 38 pregnant women with MDD will be randomized to receive sham transcranial magnetic stimulation.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active Transcranial Magnetic Simulation — Subjects will be given active TMS 5 days per week for 4 weeks for a total of 20 sessions. Each session will last approximately 10 minutes.
  Other Names: Neuronetics 2100 CRS TMS System
  Arms: Active Transcranial Magnetic Stimulation
Device: Sham Transcranial Magnetic Stimulation — Subjects will be given sham TMS 5 days per week for 4 weeks for a total of 20 sessions. The sham coil contains a shielding mechanism which diverts the magnetic field away from the patient. The sham treatment will last approximately 10 minutes.
  Other Names: The eSham System
  Arms: Sham Transcranial Magnetic Stimulation

SUMMARY:
The purpose of this study is to determine if repetitive transcranial magnetic stimulation (TMS) will alleviate symptoms of major depressive disorder (MDD) in pregnant women.

TMS uses electromagnetic impulses to encourage neurons in the brain to communicate more effectively with one another. Effective neuron communication is thought to lead to the lessening of depressive symptoms. In this study subjects require daily TMS treatment for approximately four weeks.

DETAILED DESCRIPTION:
We hypothesize that there will be a decline in the Hamilton Rating Scale for Depression (HDRS-17) scores from the beginning to end of treatment. We expect that this decrease will be significantly greater in subjects receiving active transcranial magnetic stimulation (TMS) compared to those receiving placebo TMS. Treatment response will be defined as greater than 50% reduction in HDRS-17 score.

We also hypothesize that levels of Brain Derived Neurotrophic Factor (BDNF), a protein thought to regulate mood and cognitive functioning, will increase in subjects who respond to TMS treatment. We expect BDNF levels to increase by greater than or equal to 20% in those who respond to TMS. As previously stated, TMS response will be defined as a significant decrease (50% or greater) in the HDRS-17 from baseline to end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are capable of giving written informed consent and complying with all study procedures;
* Female age 18-39 years old at date of enrollment;
* Pregnant, weeks 14-34;
* Current Depressive Symptoms;
* No change in antidepressant medication at least two weeks prior to study entry if using an antidepressant.

Exclusion Criteria:

* Any alcohol or drug abuse/dependence over the 6 months prior to study entry;
* History of a seizure disorder in subject or first degree relative;
* Anti-psychotic, lithium, or anti-convulsant medications within 2 weeks of study enrollment;
* History of known brain lesions, or severe head trauma;
* Subjects with any metallic object implanted in the skull;
* Subjects with significant cardiac disease;
* Neurological or psychiatric disorders;
* Serious medical illnesses that may compromise patient safety or study conduct;
* Currently taking a drug with known potential for fetal toxicity;
* Previous pregnancy with an adverse fetal outcome;
* Current obstetrical complications
* Actively suicidal;
* History of depression unresponsive to treatment with electroconvulsive therapy (ECT).

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, M.D., Principal Investigator — Penn Center for Women's Behavioral Wellness
Locations (1):
- Penn Center for Women's Behavioral Wellness, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Kim DR, Epperson N, Pare E, Gonzalez JM, Parry S, Thase ME, Cristancho P, Sammel MD, O'Reardon JP. An open label pilot study of transcranial magnetic stimulation for pregnant women with major depressive disorder. J Womens Health (Larchmt). 2011 Feb;20(2):255-61. doi: 10.1089/jwh.2010.2353. PMID 21314450
- [Background] Kim DR, Gonzalez J, O'Reardon JP. Pregnancy and depression: exploring a new potential treatment option. Curr Psychiatry Rep. 2009 Dec;11(6):443-6. doi: 10.1007/s11920-009-0067-0. PMID 19909665
- [Background] Kim D, O'Reardon JP. Editorial: the treatment of depression during pregnancy. Isr J Psychiatry Relat Sci. 2011;48(1):3-5. No abstract available. PMID 21572235
- [Background] Kim DR, O'Reardon JP, Epperson CN. Guidelines for the management of depression during pregnancy. Curr Psychiatry Rep. 2010 Aug;12(4):279-81. doi: 10.1007/s11920-010-0114-x. PMID 20424977
- [Background] Tjoa C, Pare E, Kim DR. Unipolar depression during pregnancy: nonpharmacologic treatment options. Womens Health (Lond). 2010 Jul;6(4):565-76. doi: 10.2217/whe.10.27. PMID 20597620
- See also: Program Website — http://www.med.upenn.edu/womenswellness/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 participants were eligible at screening to be enrolled into the treatment arm of the study.
Groups:
- Active TMS; Sham TMS: 11 pregnant women in their 2nd or 3rd trimester with a primary diagnosis of MDD
Period: Overall Study
Arm/Group | Active TMS | Sham TMS
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS | Sham TMS | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.13 (5.78) | 26.41 (5.11) | 28.27 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Scale for Depression (HDRS-17) Scores Pre- and Post- Treatment
Description: We measured changes in Hamilton Rating Scale for Depression (HDRS-17) scores from baseline to post-treatment. The HDRS-17 was administered on test days 1, 10, & 20. Scoring is based on the 17-item scale and scores of 0-7 is generally accepted to be within the normal range, indicating minimal to no depression; scores of 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale.
Time Frame: Change score from baseline to test day 20 (after 20 days of intervention)
Measure: Mean (Standard Deviation); unit: difference in units on a scale
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 11 | 11
difference in units on a scale | -13.909 (5.224) | -9.091 (7.582)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; This analysis is based on a mixed model that can handle missing data; Test type: Superiority; p = 0.003, Fisher Exact

2. Secondary Outcome: Change in Brain Derived Neurotrophic Factor (BDNF) With Active Transcranial Magnetic Simulation (TMS)
Description: We measured the levels of Brain Derived Neurotrophic Factor (BDNF) concentration across time. BDNF is a protein thought to regulate mood and cognitive functioning and research has suggested that levels may vary by severity of mood symptoms. We obtained BDNF values on test days 1 & 20.
Time Frame: Change in concentration from test day 1 to test day 20
Population: Only 4 participants from both the active and sham TMS groups were used in analysis because these participants had BDNF data at both time points. Furthermore, some samples were deemed unusable.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 4 | 4
pg/mL | 146.8775 (235.6441) | 40.0550 (131.9466)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; This analysis is based on a mixed model that can handle missing data; Test type: Superiority; p = 0.425, Regression, Logistic

ADVERSE EVENTS:
Arm/Group | Active TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11 | 0/11
Other Adverse Events (participants affected / at risk) | 4/11 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=11) | Sham TMS (N=11)
Preterm Birth (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) — Late preterm birth
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=11) | Sham TMS (N=11)
Headaches (Nervous system disorders) | 4 (17) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes